CLINICAL TRIAL: NCT06722352
Title: Preparing Assisted Living Staff to Provider Palliative Care to Residents With Dementia: Palliative Care Education in Assisted Living for Dementia Care Providers (PCEAL-DCP)
Brief Title: Palliative Care Education in Assisted Living for Dementia Care Providers (PCEAL-DCP)
Acronym: PCEAL-DCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 007811; 1RF1AG087325-01 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; End of Life; Caregiver Burden; Caregiver Burnout; Patient Participation; Self Efficacy
Keywords: end of life; palliative care; education; staff training; assisted living; dementia; dementia care; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease; Death; Caregiver Burden; Patient Participation; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two research study nurses blinded to the intervention will be trained and a rating manual provided to assist in gaining a 90% IRR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - (Experimental): Hospice nurses or social workers selected from LifePath and Suncoast Hospice organizations will train the AL interventionists on the PCEAL-DCP intervention. All hospice nurses and social workers who are facilitators will be licensed practical nurses, registered nurses or master's in social work. Prior to the intervention, the hospice facilitators will complete a four-hour workshop about the topics to cover and be trained on the protocol to follow for facilitation of the four-week PCEAL sessions so each cluster in the treatment group is trained in the same manner.
  Interventions: Behavioral: Palliative Care Training
- Control (No Intervention): Wait-listed group will receive the PCEAL-DCP curriculum after completion of the study.

INTERVENTIONS:
Behavioral: Palliative Care Training — Teaching about caring for individuals with
  Arms: Intervention -

SUMMARY:
The palliative care education in assisted living for dementia care providers (PCEAL-DCP) is a 4-week intervention (once a week for 1.5 hours, a total of 6 hours) for licensed nurses, administrators and dementia care coordinators to improve quality of dementia care outcomes

DETAILED DESCRIPTION:
This is a five-year cluster randomized trial (CRT) among 30 assisted living (AL) communities (k=30) and residents (N=450), staff (N=72) and family members (N=270) with a baseline, 3, and 6 months post-intervention follow-ups for residents, a baseline and 6-month follow-up for family and a pre- and post-test (one month), 3- and 6-month follow-up for staff and baseline AL facility information from administrators to examine dementia care outcomes.

ELIGIBILITY:
Inclusion Criteria:

The AL community eligibility criteria include a minimum of 40+ beds and provide memory care services to at least 35% of their residents, and access to hospice services from Lifepath or Suncoast Hospice. The AL size of 40+ beds is selected so we will be able to recruit a minimum of 14 residents per site, based on the power analysis for the sample size of 450 for the primary study outcome of documentation of ACP discussions.

Residents are eligible if 1) they have a dementia diagnosis confirmed by the resident's physician (physician's signature required by University of South Florida (USF) Institutional Reiew Board (IRB) in prior clinical trial) regardless of dementia severity (mild, moderate, or severe), 2) if they have been admitted to the AL in the last month, and 3) if they have a legally responsible representative who understands English.

Staff are eligible if they are currently employed with the participating study AL as a registered/licensed practical nurse, administrator, or dementia care coordinator of a memory care unit and English speaking and 21 years of age or older.

Family members are eligible if 1) they are listed as the legally responsible party in the chart records for the resident with ADRD, 2) they understand English, and 3) are at least 21 years of age or older. This could include someone related to the person, a close friend or a legal guardian who oversees the person's care and is responsible for decisions about their care.

Exclusion Criteria:

AL sites will be ineligible if 1) the are not a licensed Florida assisted living facility; 2) they have previously participated in a PCEAL-DCP clinical trial (2018-2021) to avoid possible experimental contamination effects, and 3) if no staff employed at the AL are willing to participate in the study.

Residents are ineligible if they: 1) are currently receiving hospice services because residents who receive hospice are already engaged in ACP discussions upon admission; 2) if they are discharged from assisted living to another setting (nursing home or hospital) or are admitted to hospice or have died before baseline data is collected.

Staff will be ineligible if they are not licensed nurses, administrators or dementia care coordinators of a dementia care unit or terminated/resign before baseline data is collected.

Family are ineligible if: 1) they are under 21 years of age and do not understand spoken or written English and if there is already a legal authorized representative for a resident participating in the study (one family member per resident).

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Documentation of Advance Care Planning (ACP) Discussions | Baseline, 3, and 6 months
  Resident Chart: Percent of residents in sample with documentation in chart of any discussion of ACP with residents or family, last 90 days.
  Resident Chart: Percent of residents in sample with living will, health care surrogate, durable power of attorney and do not resuscitate (DNR)s in chart. (yes/no).

SECONDARY OUTCOMES:
Hospice Use | Baseline, 3, and 6 months
  Hospice use (Secondary Outcome) Resident Chart: Percent of residents in sample admitted to hospice: Calculated based on # of residents admitted to hospice in last three months. Resident Resident Resident
  Hospice use (Secondary Outcome) Resident Chart: Percent of residents in sample admitted to hospice: Calculated based on # of residents admitted to hospice in last three months. Resident Resident Resident Percent of residents in sample admitted to hospice: Calculated based on # of residents admitted to hospice in last three months.

OTHER OUTCOMES:
Palliative Care Staff Knowledge | Baseline, 3, and 6 months
  Thompson Palliative Care Knowledge 3-items, range 1-3. (alpha = 0.81) [65]
Staff Self-Efficacy | Baseline, 3, and 6 months
  Lazenby Self-efficacy with patient- and Family-Centered Communication 12-items, range 12-60 (alpha = .91) [28]
Staff commitment | Baseline, 3, and 6 months
  Montgomery 9-items, range 9-45, (alpha =.90) [49, 54]
Staff satisfaction with org. support. | Baseline, 3, and 6 months
  Montgomery 10-items, range 10-50; (alpha = .88) [49, 54]

CONTACTS AND LOCATIONS:
Overall Officials: Debra Dobbs, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] Dobbs D, Yauk J, Vogel CE, Fanfan D, Buck H, Haley WE, Meng H. Feasibility of the Palliative Care Education in Assisted Living Intervention for Dementia Care Providers: A Cluster Randomized Trial. Gerontologist. 2024 Jan 1;64(1):gnad018. doi: 10.1093/geront/gnad018. PMID 36842068
- [Background] Bureau Y, Rodat G, Barriere H, Litoux P, Bureau B. [Cutaneous mastocytosis in adults with hepatic mastocytosis and blood monocytosis]. Bull Soc Fr Dermatol Syphiligr. 1965 Nov-Dec;72(6):850-3. No abstract available. French. PMID 5881970